CLINICAL TRIAL: NCT04452786
Title: Hormonal and Metabolic Aspects of Endoscopic Sleeve Gastroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Nora Elisabeth Hedbäck, Principal Investigator, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-19012015
Record Dates: First submitted 2020-06-19; First posted 2020-06-30 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Endoscopic Sleeve Gastroplasty; Laparoscopic Sleeve Gastrectomy; Gut Hormones; Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic sleeve gastroplasity operated patients (Other): Four test days, two days before surgery, one test day three months after surgery and one test day one year after surgery
  Interventions: Procedure: Endoscopic sleeve gastroplasty
- Laparoscopic sleeve gastrectomy operated patients (Other): Four test days, two days before surgery, one test day three months after surgery and one test day one year after surgery
  Interventions: Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Endoscopic sleeve gastroplasty — Four-hour solid mixed meal test
  Arms: Endoscopic sleeve gastroplasity operated patients
Procedure: Laparoscopic sleeve gastrectomy — Four-hour solid mixed meal test
  Arms: Laparoscopic sleeve gastrectomy operated patients

SUMMARY:
The investigators of the study want to investigate the complex interactions between glucose metabolism, food intake/weight loss, and different appetite regulating hormones after ESG in comparison with conventional laparoscopic sleeve gastrectomy (LSG).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Scheduled for endoscopic or laparoscopic sleeve at Hvidovre Hospital
* HbA1c < 48 mmol/mol before surgery, and no history of diabetes
* HbA1c < 48 mmol/mol and fasting plasma glucose < 6.1 mmol/l at inclusion
* BMI<45

Exclusion Criteria:

* Hemoglobin < 6.5 mmol/l at inclusion
* Pregnancy or breast feeding
* Medication affecting the planned examinations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Changes in ghrelin (pg/ml) | 240 minutes
  Changes in ghrelin after a solid meal test compared before and after surgery

SECONDARY OUTCOMES:
Changes in gut hormone response before and after sugery (pmol/L) | 240 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark